CLINICAL TRIAL: NCT05908448
Title: Accuracy and Precision of the True Vie I3 Continuous Glucose Monitoring System in Pediatric Patients With Type 1 Diabetes Mellitus: an Open Label, Multi-Center Trial
Brief Title: The True Vie I3 Continuous Glucose Monitoring System in Pediatric Patients With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Sinocare (Industry)
Collaborators: Atlanta Diabetes Associates (Other)
Responsible Party: Sponsor
Other Study IDs: NPI031-CIP-003F
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-02

CONDITIONS: T1DM - Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- 13-17 year old participants: 13-17 year old participants
  Interventions: Device: 13 CGM (continuous glucose monitor)
- 7-12 year old participants: 7-12 year old participants
  Interventions: Device: 13 CGM (continuous glucose monitor)
- 2-6 year old participants: 2-6 year old participants
  Interventions: Device: 13 CGM (continuous glucose monitor)

INTERVENTIONS:
Device: 13 CGM (continuous glucose monitor) — The I3 CGM consists of three main components: a Sensor Pack (Applicator-Sensor assembly), a Transmitter Pack (with Bluetooth Low Energy (BLE)) and a mobile application (I3 CGM App). The user can view their glucose data on the I3 CGM App running on a compatible mobile device.

SUMMARY:
The purpose of the investigation is to evaluate the performance of the I3 CGM in Pediatric Patients with Type 1 Diabetes Mellitus (T1DM) according to the FDA's special controls for iCGM.

DETAILED DESCRIPTION:
All participants have T1DM and will continue normal daily activities and manage their glucose as usual between clinic visits. Participants will not have access to the I3 CGM data for the management of their BG between clinic visits and will continue their usual care including CGM, if they are CGM users.

2-6 year old participants: Participants will have 2 sensors inserted in the upper buttocks by their guardian.

Participants will complete one frequent sampling clinic visit of 4 hour duration with the goal of 10-15 BG measurements analyzed using a BG meter.

For the 2-6 year olds, there are no specific fasting or other dietary requirements during the visits, participants will be provided meal choices as needed when they are hungry and meals will be served as it fits the clinic's schedule. Study staff will determine meal and insulin doses. No attempts at manipulating glucose will be made in this age group.

7-17 year old participants will attend a screening visit, an I3 CGM insertion visit, 2 clinic visits with frequent sample testing (FST) of 6 hour duration early and late in the 15 day I3 CGM sensor life. At the 2 FST clinic visits venous blood samples will be drawn for FST over 6 hours for plasma glucose determination using a Yellow Springs Instrument 2300 Stat Plus Glucose and Lactate Analyzer (YSI).

Participants will wear 3 sensors in two anatomical locations for 15 days and complete a 6 hour frequent sampling day at the beginning and the end of the sensor life.

For the 7-12 year olds, there are no specific fasting or other dietary requirements during the visits, participants will be provided meal choices as needed when they are hungry and meals will be served as it fits the clinic's schedule. Study staff will determine meal and insulin doses. No attempts at manipulating glucose will be made in this age group.

For the 13-17 year old participants, the investigative site staff will determine the participants' insulin doses and food intake and thus manipulate blood glucose to study the device over its full operating range. There will only be one glucose manipulation session during a FST visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T1DM diagnosed for at least 6 months aged 2-17 years old, inclusive.
2. Must be and have been in stable treatment regimen for at least 1 month with a multiple daily insulin dosing regimen or CSII, irrespective of delivery device(s). For this criterion, "stable treatment regimen" is considered no changes in prescribed number of insulin deliveries a day, and a change in total daily insulin dose of less than 10%.

Exclusion Criteria:

1. History of skin adhesive tolerance issues in the area of sensor placement.
2. Insulin meal dosing based on fixed dose regimens.
3. For 13-17 years old only: Absence of established correction factor for high glucose.
4. Hematocrit below 10% under the lower limit of the normal range by less than 3 month old laboratory test in history, a centrifuge or POC meter test.
5. For 7-17 year old: inadequate intravenous access on arms.
6. Participant has had a severe hypoglycemic event requiring 3rd party assistance within the past 6 months prior to enrollment.
7. Conditions which may predispose subjects to hypoglycemia including, but not limited to, thyroid disease which is not well controlled, adrenal insufficiency, high dose steroid use in recent past or planned during study, significant renal or liver disease.
8. Participant has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to enrollment.
9. Participant has a history of a seizure disorder.
10. For girls of reproductive potential: pregnancy, planned pregnancy within the study period, or unwillingness to use reliable contraception during the study period.
11. Planned MRI, CT scan or diathermia procedure for the duration of the study.
12. Any medical history of malignant melanoma or breast cancer.
13. Medical history of any other cancers within the last five years except adequately treated basal cell or squamous carcinoma of the skin, or cervical carcinoma in-situ.
14. Medical history of stroke, transitory cerebral ischemia, myocardial infarction, unstable angina or heart failure with in the past 12 months.
15. History of alcohol or drug abuse within the last year.
16. Participant has donated or lost >5% of estimated blood volume or more of their blood volume within 45 days prior to Day 0.
17. Any condition that in the opinion of the investigator may interfere successful completion of study procedures.
18. Participant is actively participating in an investigational study (e.g., drug or device) wherein he/she has received treatment from an investigational study (drug or device) in the last 2 weeks prior to Visit 1. Please note participation in observational study is acceptable.
19. Participant is a member of the research staff involved with the study.
20. Inability or unwillingness to conform to the required protocol procedures including both participant and guardian giving informed consent, and for 7-17 years old only also hypoglycemia and hyperglycemia induction.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2-17 year old patients with type 1 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Accuracy | 0-15 days
  percentage of iCGM values in the measuring range less than 70 mg/dL (3.9 mmol/l) within +/- 15 mg/dL (0.83 mmol/l) of the YSI control

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates
Locations (1):
- Atlanta Diabetes Associates, Atlanta, Georgia, United States